CLINICAL TRIAL: NCT07376824
Title: Clinical and Metabolomics Studies on the Improvement of Ovarian Reserve by Acupoint Photodynamic Therapy and Traditional Chinese Medicine Treatment
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SF2024
Record Dates: First submitted 2025-12-02; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-11

CONDITIONS: Diminished Ovarian Reserve (DOR)
Keywords: diminished ovarian reserve; Integrated Traditional Chinese and Western Clinical Medicine; Randomized controlled trial; Photodynamic Therapy; metabolomics
MeSH Terms: interventions — Medicine, Chinese Traditional; Photochemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Combination Therapy Group (Experimental): LLLT (acupoint photodynamic therapy) + Dingkun Dan Group
  Interventions: Drug: Traditional Chinese Medicine; Device: Photodynamic therapy (PDT)
- Photodynamic Therapy Group (Placebo Comparator): LLLT (acupoint photodynamic therapy) + placebo (Dingkun Dan Simulant)
  Interventions: Device: Photodynamic therapy (PDT); Drug: Placebo
- Chinese Medicine Group (Active Comparator): Dingkun Dan Monotherapy Group
  Interventions: Drug: Traditional Chinese Medicine

INTERVENTIONS:
Drug: Traditional Chinese Medicine — Dingkun Dan 7g, twice daily (bid) for 21 days per month, administered orally for 3 treatment cycles.
  Arms: Chinese Medicine Group; Combination Therapy Group
Device: Photodynamic therapy (PDT) — LLLT: The acupoint phototherapy device, with a peak wavelength of 630nm ± 20nm and an output optical power of 1-2.5mW, was used. Treatment commenced after the end of the menstrual period, once daily for 20 minutes per session, for 5 days (constituting one treatment cycle). After a 2-day interval, the next treatment cycle began, continuing until the onset of the next menstruation.
  Arms: Combination Therapy Group; Photodynamic Therapy Group
Drug: Placebo — Placebo: Simulated Dingkun Dan preparation, 7g, twice daily (bid) for 21 days per month, administered orally for 3 treatment cycles.
  Arms: Photodynamic Therapy Group

SUMMARY:
Diminished Ovarian Reserve (DOR) refers to a reduction in the number of recruitable follicles in the ovaries and/or a decline in oocyte quality. Current research on its etiology and treatment remains unsatisfactory. This study will be conducted as a single-center, prospective, parallel, randomized, controlled clinical trial in DOR patients. Eligible subjects will be randomly assigned to three groups: LLLT (acupoint photodynamic therapy) + placebo (Dingkun Dan Simulant), LLLT (acupoint photodynamic therapy) + Chinese medicine (Dingkun Dan), and Chinese medicine (Dingkun Dan) alone. Clinical data and serum metabolomics will be assessed at baseline and after the 3-month treatment.

DETAILED DESCRIPTION:
Ovarian reserve can reflect a woman's fertility and the outcomes of assisted reproductive technology. If not treated promptly, it may progress to Premature Ovarian Failure (POF) within 1 to 6 years, severely affecting a woman's physical and mental health. Studies have found that the incidence of DOR in the female population is approximately 10%, while the prevalence of DOR among infertile women is about 24%, showing an increasing trend year by year and affecting younger age groups. Extensive studies have confirmed that traditional Chinese medicine, as well as integrated traditional Chinese and Western medicine treatments, have certain therapeutic effects on DOR in clinical practice. Early intervention for DOR can improve ovarian reserve function and increase the pregnancy rate. This study will be conducted as a prospective, randomized, controlled clinical trial. Eligible subjects will be randomly assigned to three groups: Combination Therapy Group, Photodynamic Therapy Group, Chinese Medicine Group. After three months of treatment, the study will conduct clinical and metabolomics-based research on DOR patients to: (1) Clarify the role and efficacy of acupoint photodynamic therapy, both alone and in combination with Chinese medicine, in improving or enhancing the effects of traditional Chinese medicine on ovarian reserve function. (2) Explore new metabolic biomarkers for the diagnosis and efficacy evaluation of ovarian reserve function. (3) Identify the distinct metabolic pathways through which acupoint photodynamic therapy and Chinese medicine improve ovarian reserve function. (4) Establish an integrated biomarker index system for the diagnosis and treatment evaluation of DOR using acupoint photodynamic therapy and traditional Chinese medicine, and elucidate the mechanisms of action and pharmacodynamic material basis for improving ovarian reserve function.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 25 to 40 years

  * Meet the diagnostic criteria for diminished ovarian reserve (requiring at least two of the following: Basal FSH 10-25 IU/L; AMH < 1.1 ng/mL; AFC < 7) ③ Meet the diagnostic criteria for kidney deficiency syndrome in traditional Chinese medicine ④ Voluntarily participate in this study and provide written informed consent.

Exclusion Criteria:

* Organic lesions such as ovarian tumors, pituitary adenomas, endometrial tuberculosis, intrauterine adhesions or endometrial damage after abortion, as well as polycystic ovary syndrome, hyperprolactinemia, congenital adrenal hyperplasia, Cushing's syndrome, and thyroid dysfunction

  * Female infertility patients who have been treated with sex hormones in the past 3 months ③ Serious or unstable physical diseases, including liver, kidney, gastrointestinal, cardiovascular, respiratory, endocrine, neurological, immune or hematological, neurological and psychiatric systems,

    * History of substance (alcohol or drug) abuse or dependence within the past 3 months; heavy smokers (defined as those who smoke 20 or more cigarettes per day)

      * Previous allergy to the investigational drug or photosensitivity, or individuals with contraindications to Dingkun Dan ⑥ Have participated in another clinical trial of a investigational drug within the month prior to inclusion in this study (first interview) ⑦ Other conditions that, in the judgment of the investigator, may reduce the likelihood of enrollment or complicate the enrollment process, such as frequent job changes or other circumstances prone to loss to follow-up.

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in serum anti-Müllerian hormone (AMH) concentration | At 3 months after treatment initiation.
  Change in serum anti-Müllerian hormone (AMH) concentration, measured as the difference from baseline.
Change in serum follicle-stimulating hormone (FSH) concentration | At 3 months after treatment initiation.
  Change in serum follicle-stimulating hormone (FSH) concentration, measured as the difference from baseline.
Change in antral follicle count (AFC) | At 3 months after treatment initiation.
  Change in antral follicle count (AFC), measured as the difference from baseline.

SECONDARY OUTCOMES:
Change in serum concentrations of biochemical markers | At 3 months after treatment initiation.
  Changes in serum concentrations of prostaglandin E2 (PGE2), prostaglandin F2α (PGF2α), endothelin (ET), nitric oxide (NO), β-endorphin, and oxytocin (OT), measured as the change from baseline.
Change in menstrual blood loss assessed by the Pictorial Blood Loss Assessment Chart (PBAC) | At 3 months after treatment initiation.
  Change in menstrual blood loss assessed using the Pictorial Blood Loss Assessment Chart (PBAC), a validated semi-quantitative scale ranging from 0 to >500, with higher scores indicating greater menstrual blood loss, measured as the change from baseline.
Change in traditional Chinese medicine (TCM) syndrome score for menstrual disorders | At 3 months after treatment initiation.
  Change in traditional Chinese medicine (TCM) syndrome score for menstrual disorders assessed using a quantitative TCM syndrome differentiation scale for menstrual disorders, consisting of major and minor symptom items. The total score ranges from 0 to 42, with higher scores indicating greater symptom severity, measured as the change from baseline.
Change in health-related quality of life | At 3 months after treatment initiation.
  Change in health-related quality of life assessed using the 36-Item Short Form Health Survey (SF-36), a validated questionnaire with domain scores ranging from 0 to 100, where higher scores indicate better health-related quality of life, measured as the change from baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking union medical college hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No